CLINICAL TRIAL: NCT06475768
Title: The Influence of Menopausal Status on Myocardial Stiffness and Exercise Capacity Among Female Masters Endurance Athletes.
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kathryn F. Larson, Senior Associate Consultant, Cardiovascular Medicine, Mayo Clinic
Other Study IDs: 24-001460
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Myocardial Stiffness
MeSH Terms: interventions — Echocardiography, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Premenopausal Female Athletes
  Interventions: Diagnostic Test: Stress Echocardiogram; Diagnostic Test: Cardiovascular Magnetic Imaging (cMRI); Diagnostic Test: Cardiac Magnetic Resonance Elastography (cMRE)
- Postmenopausal Female Athletes
  Interventions: Diagnostic Test: Stress Echocardiogram; Diagnostic Test: Cardiovascular Magnetic Imaging (cMRI); Diagnostic Test: Cardiac Magnetic Resonance Elastography (cMRE)
- Male Athletes
  Interventions: Diagnostic Test: Stress Echocardiogram; Diagnostic Test: Cardiovascular Magnetic Imaging (cMRI); Diagnostic Test: Cardiac Magnetic Resonance Elastography (cMRE)

INTERVENTIONS:
Diagnostic Test: Stress Echocardiogram — Exercise testing via treadmill with simultaneous gas exchange analysis and pre- and post-exercise transthoracic echocardiography.
Diagnostic Test: Cardiovascular Magnetic Imaging (cMRI) — Non-invasive imaging scan used to examine function and structure of the heart
Diagnostic Test: Cardiac Magnetic Resonance Elastography (cMRE) — Non-invasive imaging scan used to measure myocardial stiffness

SUMMARY:
The purpose of this research is to study postmenopausal female masters athletes to see if they will show greater myocardial stiffness and reduced exercise capacity than premenopausal females and similarly aged male masters athletes.

ELIGIBILITY:
Inclusion Criteria:

* Longstanding history of competitive endurance athletic performance defined as >15 years of continuous athletic training for at least 7 hours per week and ongoing engagement in competitive events.

Exclusion Criteria:

* A current or prior diagnosis of cardiovascular disease as defined by the presence of structural heart disease, heart failure, symptomatic coronary artery disease, more than moderate valve disease or prior valve surgery,
* Current or recent pregnancy within 1 year
* Positive pregnancy test (study visit 1)
* Concurrent or use within 1 year of oral contraceptives or hormone replacement therapy,
* Unable to undergo a cMRI (Please refer standard clinical contraindications for MRI)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Masters athletes (40-70 yrs of age) with a longstanding history of competitive endurance athletic performance defined as >15 years of continuous athletic training for at least 7 hours per week, and ongoing engagement in competitive events, will be recruited from Mayo registry and from the local athletic community via brochures within the Dan Abraham Healthy Living Center and the Mayo Clinic Classifieds.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-10-06 (Actual); Study Completion 2025-10-06 (Actual)

PRIMARY OUTCOMES:
Myocardial stiffness | Day 14
  Myocardial stiffness will be measured by magnetic resonance elastography (kPa)

SECONDARY OUTCOMES:
Left ventricular filling pressures with exercise | Baseline
  Left ventricular filling pressures with exercise will be measured by stress echocardiography
Exercise capacity | Baseline
  Exercise capacity will be measured by stress echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Larson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No